CLINICAL TRIAL: NCT02123511
Title: A Randomized, Double-Blind Pilot Study of N-Acetylcysteine Mucoadherent Rinse Versus Placebo for Thickened Secretions and Mucositis Secondary to Chemoradiotherapy in the Management of Head and Neck Malignancies
Brief Title: Acetylcysteine Rinse in Reducing Saliva Thickness and Mucositis in Patients With Head and Neck Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC13C2; NCI-2014-00865 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Mod13-007632-07; MC13C2 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2018-12

CONDITIONS: Mucositis; Oral Complications; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Basal Cell Carcinoma of the Lip; Stage I Lymphoepithelioma of the Nasopharynx; Stage I Lymphoepithelioma of the Oropharynx; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Salivary Gland Cancer; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Nasopharynx; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Adenoid Cystic Carcinoma of the Oral Cavity; Stage II Basal Cell Carcinoma of the Lip; Stage II Lymphoepithelioma of the Nasopharynx; Stage II Lymphoepithelioma of the Oropharynx; Stage II Mucoepidermoid Carcinoma of the Oral Cavity; Stage II Salivary Gland Cancer; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Nasopharynx; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Basal Cell Carcinoma of the Lip; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Lymphoepithelioma of the Oropharynx; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVA Basal Cell Carcinoma of the Lip; Stage IVA Lymphoepithelioma of the Oropharynx; Stage IVA Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVB Basal Cell Carcinoma of the Lip; Stage IVB Lymphoepithelioma of the Oropharynx; Stage IVB Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVC Basal Cell Carcinoma of the Lip; Stage IVC Lymphoepithelioma of the Oropharynx; Stage IVC Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Mucositis; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (acetylcysteine) (Experimental): Patients receive acetylcysteine oral rinse and gargle or swish for 60 seconds then spit 5 times per day beginning within 3 days of the initiation of radiotherapy to 14 days following completion of radiotherapy.
  Interventions: Drug: acetylcysteine; Other: quality-of-life assessment; Other: questionnaire administration
- Arm II (placebo) (Placebo Comparator): Patients receive a placebo oral rinse and gargle or swish for 60 seconds and then spit 5 times per day beginning within 3 days of the initiation of radiotherapy to 14 days following completion of radiotherapy.
  Interventions: Other: placebo; Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Drug: acetylcysteine — Oral rinse
  Other Names: Airbron; Broncholysin; Brunac; N-acetylcysteine; NAC
  Arms: Arm I (acetylcysteine)
Other: placebo — Oral rinse
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies whether acetylcysteine oral rinse will lessen saliva thickness and painful mouth sores in patients with head and neck cancer undergoing radiation therapy. Side effects from radiation therapy to the head and neck, such as thickened saliva and mouth sores, may interfere with activities of daily living such as eating and drinking, and may also cause treatment to be stopped or delayed. Acetylcysteine rinse may reduce saliva thickness and mouth sores, and improve quality of life in patients with head and neck cancer undergoing radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effectiveness of N-acetylcysteine (acetylcysteine) in improving saliva viscosity (as measured by the Groningen Radiotherapy-Induced Xerostomia [GRIX]) in patients undergoing chemotherapy and radiotherapy for head and neck cancer.

SECONDARY OBJECTIVES:

I. To determine whether N-acetylcysteine (NAC) can improve other GRIX subscale for patients undergoing chemotherapy and radiotherapy for head and neck cancer.

II. To determine whether NAC can improve patient reported quality of life as measured by the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire (QLQ) Head & Neck (H&N)35.

III. To assess the adverse event profile of NAC as measured by the Common Terminology Criteria for Adverse Events (CTCAE) every week during radiation.

IV. To determine patient adherence to N-acetylcysteine mucoadherent rinse using patient reported surveys.

V. To determine the long-term benefits of N-acetylcysteine as measured by the GRIX questionnaire at 45 days and 90 days post treatment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive acetylcysteine oral rinse and gargle or swish for 60 seconds then spit 5 times per day, beginning within 3 days of the initiation of radiotherapy to 14 days following completion of radiotherapy.

ARM II: Patients receive a placebo oral rinse and gargle or swish for 60 seconds and then spit 5 times per day beginning within 3 days of the initiation of radiotherapy to 14 days following completion of radiotherapy.

After completion of study treatment, patients are followed up at 45 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of tumor of the oral cavity, oropharynx, supraglottic larynx, or nasopharynx
* Receiving concurrent chemoradiotherapy/chemobiotherapy to a minimum dose equivalent to 60 Gy in 30 fractions in the adjuvant or definitive setting
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Initiation of investigational agent =< 3 days after initiation of radiotherapy
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to return mail-in questionnaires during the observation phase of the study

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Receipt of induction chemotherapy
* Previous receipt of head and neck irradiation
* Utilization of amifostine during radiotherapy
* Greater than or equal to grade 2 dry mouth prior to chemoradiotherapy or greater than or equal to grade 2 mucositis
* Previous intolerance/adverse effect/allergy to any component of the placebo or active agent
* History of Sjogren's, lupus or scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Halyard, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - State University of New York Upstate Medical University, Syracuse, New York
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota

REFERENCES:
- [Derived] Sio TT, Blanchard MJ, Novotny PJ, Patel SH, Rwigema JM, Pederson LD, McGee LA, Gamez ME, Seeger GR, Martenson JA, Grover Y, Neben Wittich MA, Garces YI, Foote RL, Miller RC, Halyard MY. N-Acetylcysteine Rinse for Thick Secretion and Mucositis of Head and Neck Chemoradiotherapy (Alliance MC13C2): A Double-Blind Randomized Clinical Trial. Mayo Clin Proc. 2019 Sep;94(9):1814-1824. doi: 10.1016/j.mayocp.2019.03.031. Epub 2019 Aug 9. PMID 31405750

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Placebo): Patients receive a placebo oral rinse and gargle or swish for 60 seconds and then spit 5 times per day beginning within 3 days of the initiation of radiotherapy to 14 days following completion of radiotherapy.
- Arm B (Rincinol): Patients receive acetylcysteine oral rinse and gargle or swish for 60 seconds then spit 5 times per day beginning within 3 days of the initiation of radiotherapy to 14 days following completion of radiotherapy.
Period: Overall Study
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Started | 18 | 16
Eligible Patients | 17 | 15
Completed (evaluable for Primary Endpoint (AUC for GRIX Sticky Saliva Total Score)) | 16 | 12
Not Completed | 2 | 4
Not completed — Cancelled treatment | 1 | 0
Not completed — Incomplete data | 1 | 3
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients are included in this participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Placebo) | Arm B (Rincinol) | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.3) | 60.9 (10.3) | 58.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Groningen Radiotherapy-Induced Xerostomia (GRIX) Sticky Saliva Total Score Area Under the Curve (AUC)
Description: Groningen Radiotherapy-Induced Xerostomia (GRIX) sticky saliva total score Area under the curve (AUC).The GRIX questionnaire is a 14-item questionnaire with four subscales on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale. AUC will be calculated for each patient from baseline to two weeks following radiotherapy. The AUC values will be compared between the two arms using t-test (equal variance).
Time Frame: Up to 2 weeks following radiotherapy
Population: evaluable for Primary Endpoint (AUC for GRIX Sticky Saliva Total Score)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 16 | 12
score on a scale | 40.9 (23.7) | 27.2 (21.0)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.1232, t-test, 1 sided

2. Secondary Outcome: Groningen Radiotherapy-Induced Xerostomia (GRIX) Sticky Saliva Daytime Area Under the Curve (AUC)
Description: Groningen Radiotherapy-Induced Xerostomia (GRIX) sticky saliva Daytime Area under the curve (AUC).The GRIX questionnaire is a 14-item questionnaire with four subscales on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale. AUC will be calculated for each patient from baseline to two weeks following radiotherapy. The AUC values will be compared between the two arms using t-test (equal variance).
Time Frame: Up to 90 days after completion of radiation therapy
Population: evaluable for Primary Endpoint we included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 16 | 12
score on a scale | 45.2 (26.4) | 26.1 (18.7)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.0422, t-test, 1 sided

3. Secondary Outcome: Groningen Radiotherapy-Induced Xerostomia (GRIX) Sticky Saliva Nighttime Area Under the Curve (AUC).
Description: Groningen Radiotherapy-Induced Xerostomia (GRIX) sticky saliva Nighttime Area under the curve (AUC).The GRIX questionnaire is a 14-item questionnaire with four subscales on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale. AUC will be calculated for each patient from baseline to two weeks following radiotherapy. The AUC values will be compared between the two arms using t-test (equal variance).
Time Frame: Up to 90 days after completion of radiation therapy
Population: evaluable for Primary Endpoint we included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 16 | 12
score on a scale | 34.5 (22.8) | 29.1 (26.3)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.5634, t-test, 1 sided

4. Secondary Outcome: GRIX Xerostomia Daytime AUC
Description: GRIX Xerostomia Daytime AUC. The GRIX questionnaire is a 14-item questionnaire with four subscales on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale. AUC will be calculated for each patient from baseline to two weeks following radiotherapy. The AUC values will be compared between the two arms using t-test (equal variance).
Time Frame: Up to 90 days after completion of radiation therapy
Population: Patients who completed the GRIX Xerostomia Daytime at all specified time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 14 | 12
score on a scale | 44.1 (17.8) | 27.3 (17.9)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.02, t-test, 1 sided

5. Secondary Outcome: GRIX Xerostomia Nighttime AUC
Description: GRIX Xerostomia Nighttime AUC. The GRIX questionnaire is a 14-item questionnaire with four subscales on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale. AUC will be calculated for each patient from baseline to two weeks following radiotherapy. The AUC values will be compared between the two arms using t-test (equal variance).
Time Frame: Up to 90 days after completion of radiation therapy
Population: Patients who completed the GRIX Xerostomia Nighttime at all specified time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 16 | 12
score on a scale | 39.8 (16.4) | 31.3 (19.6)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.22, t-test, 1 sided

6. Secondary Outcome: GRIX Xerostiomia Total Score AUC
Description: GRIX Xerostiomia Total Score AUC. The GRIX questionnaire is a 14-item questionnaire with four subscales on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale. AUC will be calculated for each patient from baseline to two weeks following radiotherapy. The AUC values will be compared between the two arms using t-test (equal variance).
Time Frame: Up to 90 days after completion of radiation therapy
Population: Patients who completed the GRIX Xerostomia Total Score at all specified time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 14 | 12
score on a scale | 43.8 (14.7) | 28.5 (17.6)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.02, t-test, 1 sided

7. Secondary Outcome: EORTC Quality of Life Questionnaire (QLQ) H&N Pain AUC
Description: Average Area Under the Curve per assessment (aAUCpa) of QLQ H&N35 subscales including pain, swallowing, teeth, opening mouth, dry mouth, sticky saliva, senses problems, coughing, speech problems, felt ill, trouble with social contact, trouble with social eating, less sexuality, pain killers, nutritional supplements, feeding tube, weight loss, and weight gain. The QLQ H&N35 scoring algorithm was used for pain (questions 31-34) on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient and subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale.
Time Frame: Up to 90 days after completion of radiation therapy
Population: Patients who completed the QLQ H&N Pain at all specified time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 12 | 8
score on a scale | 32.4 (15.3) | 32.0 (13.9)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.95, t-test, 1 sided

8. Secondary Outcome: EORTC Quality of Life Questionnaire (QLQ) Swallowing
Description: Average Area Under the Curve per assessment (aAUCpa) of QLQ H&N35 subscales including pain, swallowing, teeth, opening mouth, dry mouth, sticky saliva, senses problems, coughing, speech problems, felt ill, trouble with social contact, trouble with social eating, less sexuality, pain killers, nutritional supplements, feeding tube, weight loss, & weight gain. The QLQ H&N35 scoring algorithm was used for swallowing (questions 35-38) on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient & subscale, the subscale values at treatment-initiation & assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale.
Time Frame: Up to 90 days after completion of radiation therapy
Population: Patients who completed the QLQ H&N Swallowing at all specified time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 10 | 8
score on a scale | 34.7 (18.8) | 22.3 (17.6)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.17, t-test, 1 sided

9. Secondary Outcome: EORTC Quality of Life Questionnaire (QLQ) H&N Sticky Saliva AUC
Description: Average Area Under the Curve per assessment (aAUCpa) of QLQ H&N35 subscales including pain, swallowing, teeth, opening mouth, dry mouth, sticky saliva, senses problems, coughing, speech problems, felt ill, trouble with social contact, trouble with social eating, less sexuality, pain killers, nutritional supplements, feeding tube, weight loss, & weight gain. The QLQ H&N35 scoring algorithm was used for sticky saliva (question 42) on 0-100 scales with higher scores representing worse symptoms. The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the end of radiotherapy. For example; for each patient & subscale, the subscale values at treatment-initiation & assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to the end of their radiotherapy are averaged to yield the aAUCpa per patient per subscale.
Time Frame: Up to 90 days after completion of radiation therapy
Population: Patients who completed the QLQ H&N Sticky Saliva at all specified time points are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 12 | 8
score on a scale | 46.3 (22.8) | 37.9 (28.5)
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.48, t-test, 1 sided

10. Secondary Outcome: Adverse Event, as Measured by the Number of Patients With a Maximum Grade of Any Adverse Event
Description: The maximum grade for each type of toxicity will be recorded for each patient. The overall adverse event rates (percentages) for adverse events are reported below.
Time Frame: Up to 90 days after completion of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
Number analyzed (Participants) | 17 | 15
Participants
  Missing | 0 | 1
  Grade 0 | 2 | 0
  Grade 1 | 3 | 5
  Grade 2 | 4 | 6
  Grade 3 | 8 | 3
Statistical Analysis 1: Comparison: Arm A (Placebo) vs Arm B (Rincinol); Test type: Superiority; p = 0.3824, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events are collected weekly during radiotherapy management visits
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed the AE form at least once. Serious AE (SAE) reports may include any secondary serious/non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm A (Placebo) | Arm B (Rincinol)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/17 | 0/16
Other Adverse Events (participants affected / at risk) | 15/17 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Placebo) (N=17) | Arm B (Rincinol) (N=16)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Placebo) (N=17) | Arm B (Rincinol) (N=16)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 1 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 11 (28) | 7 (13)
Oral hemorrhage (Gastrointestinal disorders) | 4 (10) | 2 (7)
Oral pain (Gastrointestinal disorders) | 11 (47) | 8 (31)
Creatinine increased (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes